CLINICAL TRIAL: NCT06959901
Title: Investigating the Efficacy of Mobile Health Monitoring and Self-care to Improve Obesity Outcomes in Hispanic Adolescence Populations
Brief Title: PATHS-UP Health Behavior Self-monitoring Mobile App for Adolescents
Acronym: PATHS-UP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Erica Gabrielle Soltero Ngwolo, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-55556
Record Dates: First submitted 2025-04-14; First posted 2025-05-07 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Obesity and Diabetes Mellitus, Type 2; Diabetes Prevention
Keywords: mHealth; Digital health; teen health; lifestyle intervention; mobile phone app
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile App (Experimental): Youth in the intervention will be given access to a health-based mobile phone application and a remote bluetooth scale. The app is focused on promoting health education and self-monitoring. For 30 days youth will be asked to engage with content focused on promoting healthy sleep, physical activity, and dietary habits every day. Youth will also be asked to self-monitor health behaviors using the app as it pulls in data on daily steps from the accelerometer embedded within the smartphone, information on weight from daily weigh-ins using the remote scale, sleep via weekly surveys within the app, and caloric intake using a daily food log that is powered through artificial intelligence within the app.
  Interventions: Behavioral: PATHS-UP Mobile Phone Application

INTERVENTIONS:
Behavioral: PATHS-UP Mobile Phone Application — Youth in the intervention will be given access to a health-based mobile phone application and a remote bluetooth scale. The app is focused on promoting health education and self-monitoring. For 30 days youth will be asked to engage with content focused on promoting healthy sleep, physical activity, and dietary habits every day. Youth will also be asked to self-monitor health behaviors using the app as it pulls in data on daily steps from the accelerometer embedded within the smartphone, information on weight from daily weigh-ins using the remote scale, sleep via a weekly survey within the app, and caloric intake using a daily food log that is powered through artificial intelligence within the app.

SUMMARY:
Hispanic adolescents in the U.S. are disproportionately burdened by type 2 diabetes (T2D) compared to non-Hispanic white youth (0.079% vs. 0.017%) contributing to higher rates of T2D-related vascular complications, cardiovascular disease, and mortality, among this population. Disparities in T2D are driven in part by independent, modifiable risk factors including low levels of physical activity, sleep, and poor diet. Lifestyle interventions are the cornerstone for maintaining glucose control and managing T2D. However, few studies have developed and tested lifestyle interventions for Hispanic youth with T2D. Digital health interventions that promote healthy lifestyle behaviors like physical activity, sleep, and diet, have demonstrated effectiveness among adults. Studies that use health-based smartphone applications have demonstrated preliminary efficacy for improving health-related lifestyle behaviors as these digital tools leverage behavior change techniques (e.g. self-monitoring, goal-setting, feedback) that have proven effective. Use of digital technology allows for the continuous delivery of intervention content into the home environment extending the reach of clinical care while engaging youth in a format that is age-appropriate given that today's youth are digital frontrunners. Unfortunately, while the use of digital health interventions have increased, few studies have focused on adolescents with overweight and obesity who are at high risk for T2D. The purpose of this study is to 1) develop a mobile health platform for remote and continuous monitoring of activity, sleep, and nutrition and 2) conduct a pilot study (30 days) to evaluate the efficacy of a novel digital health platform in improving obesity-related health outcomes outcomes in Hispanic adolescents (12-18 years; N=30) population.

DETAILED DESCRIPTION:
To test the feasibility and acceptability of a health-based mobile phone application the research team will recruit a sample of Hispanic adolescents (12-18 years; N=30) with overweight and obesity. Once informed consent and youth assent have been collected, youth will be enrolled into the intervention. Investigators will leverage an existing digital monitoring platform consisting of a Bluetooth-enabled weight scale and the mobile health app developed through Apple iOS which provides advanced activity and sleep tracking features, visualizations and trends, and self-reporting functionality. This interface integrates data from the accelerometer embedded within the participant's own smartphone. This accelerometer integrates data including steps and physical activity minutes into the app. Users do not need to sign any agreements with apple or any end user licenses. All data obtained through the app is transmitted to the digital monitoring platform before it is integrated into a REDCap database. Youth will be provided with a remote bluetooth enabled scale which will transmit data into the digital platform. The app provides youth with an AI enabled component to log their daily diet as well as a weekly survey to assess sleep.

A longitudinal, pre-post design will be used to test the 30-day intervention. The investigators will leverage existing collaborations with the Department of Endocrinology at Texas Children's Hospital and an existing network of physicians within the Texas Children's Health Plan and Harris Health Pediatric Clinics. Study flyers will be placed in waiting and exam rooms and physicians in participating clinics will be encouraged to refer eligible patients to the study. The research team will also attend community-wide events such as back to school fairs and food drives at partnering community-based organizations (e.g. Baker Ripley) where the research team will pass out flyers and share study information for attendees. The research team also have a sign up sheet where interested participants can leave their contact information if they would like to receive more information about the study. Lastly, the Children's Nutrition Research Center maintains a volunteer participant registry, which includes youth who have expressed interest in participating in future research projects. Participants within the registry who are eligible will be invited via a phone call to participate in this study. These participants have consented to be contacted for future projects. The research team will also send a text message to interested participants who have consented through the registry or have volunteered their contact information at community events. This text will share a brief information video in English or Spanish to generate interest in the study.

If participants agree to join the study, they will receive information and parental consent and child assent will be obtained prior to any study procedures. Once they join the study, participants will receive an IndieHealth Bluetooth-enabled weight scale and a customized mobile health app and will be asked to conduct daily self-measurement of weight, complete daily educational tasks, and log meals for 30 days. Participants will receive instructions explaining how the accelerometer embedded within their phone will be used to integrate step and sleep data into the health app. Daily motivational and persuasive messages will be sent to participants to assist them in increasing their activity, sleep, and dietary habits towards the recommended national guidelines. Youth will also receive prompts to self-monitor their health behaviors. The messages and content that youth will receive are theory-informed and were previously developed with youth and research experts to ensure that they are theoretically adherent, culturally, and age appropriate.

Feasibility will be examined using research notes and careful documentation of recruitment, data collection, technical issues, engagement, and satisfaction. The acceptability, utility, and engagement with the mobile health platform will be measured using a study-specific, process evaluation questionnaire. This will provide information on the availability of high-risk youth in community clinics willing to participate in a digital health program and the ability to recruit, retain, and engage this population. Careful documentation of technical issues will speak to the feasibility of developing and implementing this type of technology for health promotion and disease prevention purposes.

In addition to feasibility, several outcomes will be assessed including weight, average steps/day, average minutes of sleep/night, and dietary intake as collected through the mobile health app. A remote scale will be used to measure weight, and a self-reported fat, fruit, and vegetable screener (National Cancer Institute) to assess dietary intake. Baseline and post-intervention assessments will be conducted and will consist of a demographic survey to be completed by parents. Motivation for exercise will be measured using a 9-item survey, which has shown acceptable validity and reliability among youth. Following the intervention, youth will be asked to complete a system usability scale to understand the acceptability and feasibility of the app and program from the perspective of the participant.

To further assess acceptability, an exit interview will be conducted with a subsample of participants (N=15) to evaluate the experience and identify barriers and opportunities for further redesigns. This information will also provide guidance on the acceptability of this strategy among this age and ethnic subgroup. In-depth interviews be conducted via a dedicated study line. They will be audio-recorded, transcribed, coded by two trained, independent coders, and qualitatively analyzed using NVivo version 9. Thematic content analysis will be used to identify emergent themes to adapt existing text messages. App related data (weight, steps, sleep, diet) will be monitored including engagement metrics (e.g. participant logins, app usage) and any data transmitted through the app including the food diary, step count, and weight data. All data will be de-identified and will only include a unique participant identifier in the form of a numerical number.

All surveys and assessments will be conducted remotely using secure links generated through REDCap.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Hispanic or Latino
* 12-18 years
* BMI% in the 85th-95th range,
* Owns their own iphone

Exclusion Criteria:

* Currently enrolled in a health program
* Diagnosed with T2D
* Present with a disease or condition that would prevent one from engaging in activity

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Recruitment | From enrollment to the end of the 30 day study.
  The rate of recruitment will be assessed to determine the feasibility of the research team's ability to recruit the target sample (N=30).
Feasibility of Technology | through study completion, an average of 30 days
  The number of technical issues reported by participants or the research team will be documented throughout the intervention.
Usability | At the end of the 30 day study.
  The system usability scale will be used to assess feasibility. Scores using this tool range from 0 to 100, with a higher score will indicating higher usability.
Acceptability | At the end of the 30 day study.
  Acceptability will be assessed using an exit survey. The research team will use a Likert scale to assess the acceptability of various components of the study including the mobile phone app interface, content, etc. A higher score will indicate greater satisfaction.
Acceptability | at the end of the 30 day study
  To assess acceptability, the research team will also use an exit interview to gather more in-depth perspectives on the mobile phone application, the content, and the participant's experience using the app to improve health behaviors. These interviews will be analyzed using thematic content analysis.

SECONDARY OUTCOMES:
Health beliefs | From enrollment to the end of the 30 day study.
  The health beliefs model survey will be used to assess how youth perceive their susceptibility to a health condition and the benefits of taking action, and the barriers to taking action.
Autonomous Motivation | From enrollment to the end of the 30 day study.
  A survey will be used to assess the degree to which the desire to change health behaviors is autonomously motivated. A higher score will indicate higher reported autonomous motivation.
Diet | From enrollment to the end of the 30 day study.
  Fruit & vegetable intake, fat intake, and sugar sweetened beverage intake will be assessed using the NCI diet screener.
Physical activity | From enrollment to the end of the 30 day study.
  Physical activity will be assessed using the accelerometer embedded within the participants smartphone to assess days/steps.

OTHER OUTCOMES:
Sleep | baseline, weekly through the 30 day intervention, and at post-intervention
  Self-reported survey on average minutes of sleep per night and self-rated sleep quality measured on a Likert scale of 1-5, with 5 being great sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We will share anonymous data through our institutional data registry.